CLINICAL TRIAL: NCT02048449
Title: Inter-rater Reliability of the Reflux Finding Score Based on Endoscopic Laryngeal Findings in the Diagnosis of Laryngopharyngeal Reflux Disease
Brief Title: Inter-rater Reliability of the Reflux Finding Score Among Gastroenterologists
Status: Completed | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Yeonsoo Kim, Assistant professor, Chuncheon Sacred Heart Hospital
Other Study IDs: ChuncheonSHH 2013
Record Dates: First submitted 2014-01-21; First posted 2014-01-29 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Laryngitis; Reflux
Keywords: Reflux finding score, interrater reliability
MeSH Terms: conditions — Laryngitis; Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Title:

Inter-rater reliability of the reflux finding score based on endoscopic laryngeal findings in the diagnosis of laryngopharyngeal reflux disease

Participants:

Voluntary participants after invitation among members (a total of about 40 gastroenterologists) of Gangwon Branch of Korean Society of Gastrointestinal Endoscopy and an otorhinolaryngologist

Primary endpoint:

Interrater reliability (Kappa coefficient) on the sum of reflux finding score more than 7 points between an otorhinolaryngologist and gastroenterologists (7 points means the cut-off value for the diagnosis of laryngopharyngeal reflux disease)

Secondary endpoint:

Agreement (%) on 8 items of reflux finding score for laryngopharygeal reflux among gastroenterologists

DETAILED DESCRIPTION:
Study Design

1. Recruitment of doctor participants: introduction by e-mail
2. Education on reflux finding score - standardized materials (instructional video)
3. PRETEST (15 pictures) / feedback (at-a-glance assessment format)
4. TEST 1 (50 pictures) - Acess format including 8 items at each pictures
5. Feedback education (individualized intruction of an otorhinolaryngologist)
6. TEST 2 (50 pictures) - Acess format including 8 items at each pictures
7. Test-Retest reliability - repeat Test 2 with 1 week interval (Participants should take retest of TEST 2 with the concealment of the answer)
8. Analysis

ELIGIBILITY:
Inclusion Criteria:

* Participants: Gastroenterologists (GI specialists) or trainees /
* Pictures: Endoscopic laryngeal pictures with good quality

Exclusion Criteria:

* Participants: Major other than gastroenterology /
* Pictures: Endoscopic laryngeal pictures without good quality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: not appliable
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Cohen's kappa coefficient | 5 months
  Cohen's Kappa coefficient based on the sum of reflux finding scores (7 points or more than 7) for the diagnosis of laryngopharyngeal reflux disease between an otorhinolaryngologist (reference) and participant gastroenterologists

SECONDARY OUTCOMES:
Agreement (%) at each item out of 8 items of reflux finding score | 5 months
  Agreement (%) at each item out of 8 items (subglottic edema, ventricular obliteration, laryngeal erythema, vocal cord edema, diffuse laryngeal edema, posterior commissure hypertrophy, laryngeal granuloma, thick endolaryngeal mucus) of reflux finding score

CONTACTS AND LOCATIONS:
Overall Officials: Dong Kyu Kim, MD, Study Director — Assistant professor, ENT department, Chuncheon Sacred Heart Hospital